CLINICAL TRIAL: NCT04798820
Title: A Randomized Clinical Trial of Simplified Dietary Education Versus Intensive Dietary Education on Nutritional Status After Gastrectomy
Brief Title: The Effect of Intensive Dietary Education on Nutritional Status After Gastrectomy(SING)
Acronym: SING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Moon Bae, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SMC 2020-11-016-002
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Gastrectomy
Keywords: gastric cancer; gastrectomy; dietary education; nutritional status
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Simplified dietary education(SE) versus Intensive dietary education(IE)
  1. Subtotal gastrectomy group (n=258)
  2. Total gastrectomy group (n=100)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SE-STG (Active Comparator): simplified dietary education arm in subtotal gastrectomy group.
  Interventions: Other: Dietary education(nutritional counselling)
- IE-STG (Active Comparator): intensive dietary education arm in subtotal gastrectomy group
  Interventions: Other: Dietary education(nutritional counselling)
- SE-TG (Active Comparator): simplified dietary education arm in total gastrectomy group.
  Interventions: Other: Dietary education(nutritional counselling)
- IE-TG (Active Comparator): intensive dietary education arm in total gastrectomy group
  Interventions: Other: Dietary education(nutritional counselling)

INTERVENTIONS:
Other: Dietary education(nutritional counselling) — Dietary education provided to gastrectomy patients by dietitian.

SUMMARY:
Radical gastrectomy has been known as the most effective treatment of curable gastric cancer.However, there is a high risk of malnutrition and weight loss after a gastrectomy which may be attributed to inadequate oral consumption, malabsorption and loss of the reservoir function of the stomach.Weight loss has been regarded as an independent risk factor for postoperative mortality and morbidity and It is also closely associated with a quality of life after surgery. No specific surgical technique has been proved to be effective in reducing postoperative weight loss and it seems like that dietary education and consultation is the best way to minimize weight loss in gastrectomy patients in clinical setting. In this regard, the investigators performed a retrospective pilot study to identify the effect of routinely performed (simplified) dietary education on nutritional status after gastrectomy, but it revealed that the effect of simplified dietary education on weight loss was not clear and the result implies that more intensive dietary education may be necessary after gastrectomy. The aim of this randomized controlled trial (RCT) is to elucidate the effect of intensive dietary education on nutritional status after gastrectomy in comparison with simplified dietary education.

DETAILED DESCRIPTION:
Subject 1: subtotal gastrectomy group

subject 2: total gastrectomy group

Objectives:

Primary objective: to evaluate Weight loss difference of simplified dietary education(SE) versus intensive dietary education(IE) for patients after undergoing a gastrectomy

Primary endpoint: Superiority of weight loss difference (%) of IE group between post op 1mo and 12mo

Secondary objectives:

weight loss(%) of each subgroup, nutritional parameters (PG-SGA), Calrorie intake & dietary habits, albumin, hemoglobin, iron panel (TIBC, ferritin), Absolute lymphocyte count(ALC), vit B12, homocysteine, quality of life(QOL) change

1. Nutritional parameters (PG-SGA)
2. the amount of calorie intake (Kcal, protein) & dietary habits
3. Albumin (g/dL)
4. Hemoglobin (g/dL)
5. Iron panel [TIBC (μg/dL), Ferritin (ng/mL)]
6. Absolute lymphocyte count (ALC) (10^3/μL)
7. Vitamin B12 (pg/mL)
8. Homocysteine (μmol/L)
9. Quality of life of the patients in terms of European quality of life questionnaire (EQ-5D)

ELIGIBILITY:
Inclusion Criteria:

* histologically proven primary gastric adenocarcinoma,
* T1N0, T1N1, T2N0, which are assessed by computed tomography (CT) scan (AJCC 8th classification) and intraoperative surgical staging
* location of primary tumor; antrum, or angle, , lower body or mid body of the stomach
* No evidence of other distant metastasis,
* age ≥ 20 year old, ≤ 75 year old
* no prior or posterior treatment of chemotherapy or radiation therapy against any other malignancies
* adequate organ functions defined as indicated below:

  1. WBC count: 3000/mm3 ~12,000/mm3,
  2. > serum Hemoglobin 8.0 g/dL
  3. > serum Platelet 100 000/mm3,
  4. < serum AST 100 IU/L,
  5. <serum ALT 100 IU/L,
  6. < Total Bilirubin 2.0 mg/dL,
* written signed informed consent

Exclusion Criteria:

* active double cancer (synchronous double cancer and metachronous double cancer within five disease-free years), excluding carcinoma in situ (lesions equal to intraepithelial or intramucosal cancer),
* gastric remnant cancer
* ≥T3, T4 in surgical staging before resection
* N2 or more (number of metastatic lymph nodes ≥3) in CT scan
* histologically rare variants in World Health Organization (WHO) Classification such as Adenosquamous, Hepatoid, Squamous cell, Undifferentiated, neuroendocrine carcinoma and others
* pregnant or breast-feeding women,
* mental disorder(diagnosed with mental disorder on medical record),
* unstable angina or myocardial infarction within 6 months of the trial,
* unstable hypertension,
* diabetes mellitus on insulin,
* severe respiratory disease requiring continuous oxygen therapy,
* previous upper abdominal surgery except laparoscopic cholecystectomy,
* surgical complication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative weight change at immediate postoperative period in SE and IE groups. | preoperative, immediate postoperative
  comparison of weight change between the two groups after surgery
Change from preoperative weight change at postoperaive 1 month in SE and IE groups. | preoperative, postoperative 1 month
  comparison of weight change between the two groups after surgery
Change from preoperative weight change at postoperaive 3 months in SE and IE groups. | preoperative, postoperative 3 months
  comparison of weight change between the two groups after surgery
Change from preoperative weight change at postoperaive 6 months in SE and IE groups. | preoperative, postoperative 6 months
  comparison of weight change between the two groups after surgery
Change from preoperative weight change at postoperaive 12 months in SE and IE groups. | preoperative, postoperative 12 months
  comparison of weight change between the two groups after surgery
Change from preoperative weight change at postoperaive 18 months in SE and IE groups. | preoperative, postoperative 18 months
  comparison of weight change between the two groups after surgery

SECONDARY OUTCOMES:
Nutritional parameters | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  measured by Patient-Generated Subjective Global Assessment (PG-SGA; rating A,B,C)
24hrs dietary recall | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  calculating kcal & protein intake by 24hrs dietary recall (questionnaire)
dietary habits | preoperative, immediate postoperative, postoperative 1 months, 3 months, 6months, 12 months, 18 months
  number of meals, eating speed (questionnaire)
Albumin | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  g/dL
Hemoglobin | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  g/dL
Total iron binding capacity (TIBC) | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  μg/dL
Ferritin | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  ng/mL
Absolute lymphocyte count (ALC) | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  10^3/μL
Vitamin B12 | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  pg/mL
Homocysteine | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  μmol/L
Quality of life of the patients | preoperative, immediate postoperative, postoperative 1 month, 3 months, 6months, 12 months, 18 months
  European quality of life questionnaire (EQ-5D); the descriptive system which comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems (labelled 1-3).

CONTACTS AND LOCATIONS:
Overall Officials: Aron Lee, RD, Study Director — Samsung Medical Center; Bo Ram Park, Ph.D., Study Director — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee AR, Bae JM, Choi MG, An JY, Kim EM, Park B. Nutritional Counseling for Patients With Gastric Cancer After Subtotal Gastrectomy: A Randomized Clinical Trial. J Gastric Cancer. 2025 Oct;25(4):593-604. doi: 10.5230/jgc.2025.25.e43. PMID 41093778

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04798820/SAP_001.pdf